CLINICAL TRIAL: NCT02027259
Title: Behavioral Activation Therapy for Both Depression and Diabetes Vs. Diabetes Alone Delivered Via Group Visits
Acronym: BA-MEDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracey H. Taveira, Tracey H. Taveira, Pharm.D., CDOE, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12CRP9840018
Record Dates: First submitted 2013-11-12; First posted 2014-01-06 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; Depression
Keywords: Diabetes; Depression; Group
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group visits with behavioral activation (Experimental): Group visits with behavioral activation (BA) will consist of 4 weekly group visits of 2-hour duration followed by monthly booster group visits for 6 months to prevent relapse.
  Interventions: Behavioral: Behavioral activation (BA)
- Standard group visits (No Intervention): Standard group visits will consist of 4 weekly group visits of 2-hour duration followed by monthly booster group visits for 6 months to prevent relapse.

INTERVENTIONS:
Behavioral: Behavioral activation (BA) — The addition of Behavioral activation (BA) to our group visits in patients with DM and depression will consist of 4 weekly group visits of 2-hour duration followed by monthly booster group visits for 6 months to prevent relapse.
  Other Names: BA MEDIC
  Arms: Group visits with behavioral activation

SUMMARY:
The purpose of this study is to determine whether group visits with added behavioral activation (BA) for depression will have a greater clinical impact than our standard group visits without BA for depression in reducing the risk of future coronary events as measured by the United Kingdom Prospective Diabetes Study (UKPDS) risk engine and depression symptoms as measured by Patient Health Questionnaire-9 (PHQ-9) after 6 months.

DETAILED DESCRIPTION:
BACKGROUND Nearly 33% of the 24.5 million people in the US with diabetes mellitus (DM) have co-morbid depression. Since 65% of patients with DM die from cardiovascular disease (CVD), concomitant control of CVD risk factors along with glycemic control is crucial to prevent adverse outcomes. However, co-morbid depression makes DM and CVD risk factors harder to control. We demonstrated that a pharmacist-led group visit model consisting of: 1) pharmacotherapy management for DM, hyperlipidemia and hypertension, 2) self-management education, 3) case management and 4) behavioral strategies for DM and CVD self-care behaviors, was more efficacious in improving hyperglycemia and CVD risk factors compared to standard primary care controls in a general DM population and also for patients with DM and co-morbid depression. For participants with DM and depression there was also a non-significant trend toward improvement in depression despite the lack of depression treatment.

OBJECTIVE: Our objective is to determine whether group visits with added behavioral activation (BA) for depression (cases) will have a greater clinical impact than our standard group visits without BA for depression (active control) in reducing the risk of future coronary events as measured by the United Kingdom Prospective Diabetes Study (UKPDS) risk engine and depression symptoms as measured by Patient Health Questionnaire-9 (PHQ-9) after 6 months.

RESEARCH PLAN/METHODS: The goal is to conduct a randomized-controlled pilot trial (n=25 in each arm) to evaluate the clinical effect of added BA to our group intervention in patients with DM and depression who have a Hemoglobin A1c>=8% and a PHQ-9 depression score >=10 and at least one additional CVD risk factor such as tobacco use, hyperlipidemia or hypertension not at American Heart Association and American Diabetes Association guideline recommended goals. The interventions in both arms will consist of 4 weekly group visits of 2-hour duration followed by monthly booster group visits for 6 months to prevent relapse.

The primary aims are:

* 1) To examine the effects of our group visit model with and without added BA therapy on the 10-year UKPDS coronary event risk, and PHQ-9 depression scores after 6 months
* 2) To examine the acceptability and adherence to our group visit model with and without added BA therapy by way of focus groups and attendance

The secondary aim is

* 1) To explore mediating factors of our group visit model with added BA therapy that are associated with improvement in CVD risk and depression

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Clinical diagnosis of depression
* PHQ-9 score ≥10 for depressive symptoms
* >= 18 years old
* a most recent HbA1c ≥8.0% within the previous 12 months in the chart; and
* have 1 or more of the following modifiable CVD risk factors not at target goals, defined as:
* current smoker (any cigarette smoking <30 days),
* blood pressure >130/80 mm Hg, documented at least twice in the last 6 months
* LDL cholesterol >100 mg/dL within the last 12 months.

Exclusion Criteria:

* Inability to attend the group sessions
* active psychosis of any type or organic brain injury that precludes DM self- care
* type 1 diabetes as documented in the medical chart
* pregnancy
* actively suicidal and /or
* end-stage medical illness (e.g. metastatic cancer, awaiting organ transplant)
* Patients currently enrolled in DM group programs that include medication titration within the group setting would not be eligible due to co- intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01-19 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
Change in 10-year UKPDS coronary event risk and PHQ-9 depression scores. | Change from baseline in 10-year UKPDS coronary event risk and PHQ-9 depression scores at 6 months..
  To examine the effects of our group visit model with and without added BA therapy on the 10-year UKPDS coronary event risk, and PHQ-9 depression scores after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey H Taveira, Pharm.D., Principal Investigator — Providence VAMC
Locations (1):
- Providence VAMC, Providence, Rhode Island, United States